CLINICAL TRIAL: NCT05694689
Title: Randomized Trial of Enteral Vitamin D Supplementation in Infants < 28 Weeks Gestational Age or <1000 Grams Birth Weight
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Maria del Mar Romero López, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB # 22-0217
Record Dates: First submitted 2023-01-11; First posted 2023-01-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-06

CONDITIONS: Vitamin D Deficiency
Keywords: Premature infant; Vitamin D
MeSH Terms: conditions — Vitamin D Deficiency; Premature Birth | interventions — Saline Solution; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care plus placebo (Active Comparator): Infants will receive placebo (normal saline) in the first 28 days after birth. Co-interventions will be unaffected and provided based on the judgment of the attending neonatal faculty and NICU policies and routine practices.
  Interventions: Dietary Supplement: Placebo; Other: Usual Care
- Usual care plus vitamin D supplementation (Experimental): Infants will receive cholecalciferol 800 IU/day in the first 28 days after birth, given enterally four times per day (0.5mL per dose = 200 IU) until the infant is provided 400 IU/day. At that point the study cholecalciferol will be reduced to 400 IU/day for a total supplementation of 800 IU/day.
  Interventions: Dietary Supplement: 800 IU/day vitamin D supplementation with feedings in the first 28 days after birth; Other: Usual Care

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo is normal saline, given in the first 28 days after birth, prepared to have the same volume and appearance as vitamin D, which is a clear odorless solution.
  Other Names: Normal saline
  Arms: Usual care plus placebo
Dietary Supplement: 800 IU/day vitamin D supplementation with feedings in the first 28 days after birth — 800 IU/day Vitamin D supplementation until 400 IU/ day are provided as part of usual care. At that point the intervention becomes a supplement of 400 IU/day above that given with usual care. In this way all infants in the intervention group receive 800 IU/day of vitamin D total supplementation in the first 28 days after birth with feedings.
  Other Names: Cholecalciferol
  Arms: Usual care plus vitamin D supplementation
Other: Usual Care — Co-interventions will be unaffected and provided based on the judgment of the attending neonatal faculty and NICU policies and routine practices

SUMMARY:
The objective of the study is to compare supplementation with vitamin D at 800 IU/day to usual care for the first 28 days after birth with respect to 25 (OH) vitamin D levels and indicators of likely or plausible effects of vitamin D supplementation on the function or structure of the lung, bones, immune system, and brain in extremely premature (EP) infants who are <28 weeks gestational age (GA) or <1000 grams of birth weight (BW). The study results will be analyzed as intention to treat Bayesian analyses (Frequentist analyses will also be performed).

ELIGIBILITY:
Inclusion Criteria:

* Infants born at < 28 weeks gestational age (GA) or <1000 grams birth weight (BW)
* Inborn
* Informed written consent in an Institutional Review Board (IRB)-approved manner

Exclusion Criteria:

* GA >32 weeks regardless of birth weight (BW)
* Any major congenital anomaly
* An known congenital nonbacterial infection
* Prenatal diagnosis of disorders that affect vitamin D absorption (e.g, cystic fibrosis)
* Such severe illness or immaturity that the attending neonatologist judges intensive care to be unjustified.

Ages: 24 Hours to 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
25-hydroxyvitamin D (25[OH]D) level | about 28 days after birth

SECONDARY OUTCOMES:
25-hydroxyvitamin D (25[OH]D) level | 36 weeks after birth
Type of respiratory support required at 36 weeks postmenstrual age | 36 weeks postmenstrual age (or at the time of discharge home if earlier)
  Data will be reported categorically as:
  * Number of participants who survive without respiratory support
  * Number of participants who survive with nasal cannula at ≤ 2 liters (L)/minute
  * Number of participants who survive with nasal cannula >2 L/minute or noninvasive positive airway pressure
  * Number of participants who survive with invasive mechanical ventilation
  * Number of participants who die
Length of Hospital stay | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of participants who are still on respiratory support | 22 to 26 months corrected age
  Respiratory support includes supplemental oxygen and positive pressure ventilation.
Number of days of supplemental oxygen | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of days of mechanical ventilation | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of days of positive pressure support | from time of birth to time of discharge (about 0 to 60 weeks after birth)
Number of participants who receive steroid treatment to decrease respiratory support | from baseline to 36 weeks postmenstrual age
Number of participants with pulmonary hypertension | 36 weeks postmenstrual age
Number of participants with wheezing | 2 years
Weight as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 28 days of life
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Weight as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 36 weeks postmenstrual age
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Weight as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 2 years
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Length as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 28 days of life
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Length as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 36 weeks postmenstrual age
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Length as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 2 years
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Head circumference as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 28 days of life
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Head circumference as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 36 weeks postmenstrual age
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Head circumference as assessed by sex-specific Z-score on the Fenton 2013 Growth Calculator | 2 years
  Z-scores range from -4 standard deviations to +4 standard deviations. A higher Z-score indicates a better outcome.
Number of participants with any fractures | from baseline to 36 weeks postmenstrual age
Number of participants with hospital-acquired sepsis | from day 3 after birth to the time of discharge (which is 0 to 60 weeks after birth)
Calcium level | 0 to 36 weeks postmenstrual age
Phosphorus level | 0 to 36 weeks postmenstrual age
Alkaline phosphatase level | 0 to 36 weeks postmenstrual age
Neurodevelopment as assessed by the Bayley-IV Scale of Infant and Toddler Development (Cognitive composite score) | 2 years
  Cognitive composite score ranges from 40 to 160, with a higher score indicating a better outcome.
Neurodevelopment as assessed by the Bayley-IV Scale of Infant and Toddler Development (Language composite score) | 2 years
  Language composite score ranges from 40 to 160, with a higher score indicating a better outcome.
Neurodevelopment as assessed by the Bayley-IV Scale of Infant and Toddler Development (Motor composite score) | 2 years
  Motor composite score ranges from 40 to 160, with a higher score indicating a better outcome.
Number of participants with neurodevelopmental impairment (NDI) | 2 years
Number of participants who die or have a morbidity | 36 weeks postmenstrual age
  Morbidities include retinopathy of prematurity (ROP), intraventricular hemorrhage (IVH), bronchopulmonary dysplasia (BPD), neurodevelopmental impairment (NDI), necrotizing enterocolitis (NEC), and patent ductus arteriosus (PDA).
Vitamin D status as indicated by serum concentration of 24,25(OH)2D3 as assessed by Liquid Chromatography with tandem mass spectrometry (LC-MS/MS) | about 28 days after birth
Vitamin D status as indicated by serum concentration of 24,25(OH)2D3 as assessed by LC-MS/MS | 36 weeks postmenstrual age
Vitamin D status as indicated by serum concentration of 3-epi-25(OH)D3 as assessed by LC-MS/MS | about 28 days after birth
Vitamin D status as indicated by serum concentration of 3-epi-25(OH)D3 as assessed by LC-MS/MS | 36 weeks postmenstrual age
Vitamin D status as indicated by serum concentration of 25(OH)D3 as assessed by LC-MS/MS | about 28 days after birth
Vitamin D status as indicated by serum concentration of 25(OH)D3 as assessed by LC-MS/MS | 36 weeks postmenstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Jain, MD, Principal Investigator — The University of Texas Medical Branch
Locations (1):
- The University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No